CLINICAL TRIAL: NCT01370005
Title: A Phase III Randomised, Double-blind, Placebo-controlled, Parallel Group, Efficacy and Safety Study of BI 10773 (10 mg, 25 mg) Administered Orally, Once Daily Over 12 Weeks in Hypertensive Patients With Type 2 Diabetes Mellitus
Brief Title: 12 Week Efficacy and Safety Study of Empagliflozin (BI 10773) in Hypertensive Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1245.48; 2011-000347-25 (EudraCT Number: EudraCT)
Record Dates: First submitted 2011-06-08; First posted 2011-06-09 (Estimated); Results first posted 2014-06-17 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-01

CONDITIONS: Diabetes Mellitus, Type 2; Hypertension
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension | interventions — empagliflozin

ARMS (3):
- BI 10773 low dose (Experimental): BI 10773 low dose once daily
  Interventions: Drug: Placebo; Drug: BI 10773
- BI 10773 high dose (Experimental): BI 10773 high dose once daily
  Interventions: Drug: BI 10773; Drug: Placebo
- Placebo (Placebo Comparator): Placebo tablets matching BI 10773
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo matching BI 10773 low dose
  Arms: BI 10773 low dose
Drug: BI 10773 — BI 10773 high dose once daily
  Arms: BI 10773 high dose
Drug: Placebo — Placebo matching BI 10773 low dose
  Arms: Placebo
Drug: BI 10773 — BI 10773 low dose once daily
  Arms: BI 10773 low dose
Drug: Placebo — Placebo matching BI 10773 high dose
  Arms: BI 10773 high dose
Drug: Placebo — Placebo matching BI 10773 high dose
  Arms: Placebo

SUMMARY:
This trial will evaluate safety and efficacy of BI 10773 in hypertensive patients with type 2 diabetes. Since hyperglycaemia and hypertension are key risk factors for both micro- and macrovascular complications, assessment of both glucose and blood pressure lowering effects of BI 10773 in hypertensive patients with type 2 diabetes could provide clinically highly relevant, new information for the use of BI 10773

ELIGIBILITY:
Inclusion criteria:

1. Patients >=18 years with type 2 diabetes
2. HbA1c of >= 7.0% (53 mmol/mol) and =< 10% (86 mmol/mol)
3. Mean seated systolic blood pressure 130-159 mmHg and diastolic blood pressure 80-99 mmHg

Exclusion criteria:

1. Uncontrolled hyperglycaemia with a glucose level >240 mg/dl (>13.3 mmol/L) after an overnight fast before randomization
2. Known or suspected secondary hypertension
3. Acute coronary syndrome (non-STEMI, STEMI and unstable angina pectoris), stroke or transient ischemic attack within 3 months prior to informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 825 (Actual)
Dates: Start 2011-06; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (120):
- United States (35):
  - 1245.48.10024 Boehringer Ingelheim Investigational Site, Huntsville, Alabama
  - 1245.48.10002 Boehringer Ingelheim Investigational Site, Phoenix, Arizona
  - 1245.48.10014 Boehringer Ingelheim Investigational Site, Lincoln, California
  - 1245.48.10030 Boehringer Ingelheim Investigational Site, Long Beach, California
  - 1245.48.10033 Boehringer Ingelheim Investigational Site, Long Beach, California
  - 1245.48.10027 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 1245.48.10041 Boehringer Ingelheim Investigational Site, Tustin, California
  - 1245.48.10039 Boehringer Ingelheim Investigational Site, West Hills, California
  - 1245.48.10008 Boehringer Ingelheim Investigational Site, Davie, Florida
  - 1245.48.10025 Boehringer Ingelheim Investigational Site, Edgewater, Florida
  - 1245.48.10001 Boehringer Ingelheim Investigational Site, Jacksonville, Florida
  - 1245.48.10016 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 1245.48.10035 Boehringer Ingelheim Investigational Site, Palm Harbor, Florida
  - 1245.48.10018 Boehringer Ingelheim Investigational Site, Pensacola, Florida
  - 1245.48.10032 Boehringer Ingelheim Investigational Site, Pinellas Park, Florida
  - 1245.48.10012 Boehringer Ingelheim Investigational Site, Marietta, Georgia
  - 1245.48.10011 Boehringer Ingelheim Investigational Site, Addison, Illinois
  - 1245.48.10019 Boehringer Ingelheim Investigational Site, Arlington Heights, Illinois
  - 1245.48.10022 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 1245.48.10017 Boehringer Ingelheim Investigational Site, Wichita, Kansas
  - 1245.48.10010 Boehringer Ingelheim Investigational Site, Albuquerque, New Mexico
  - 1245.48.10036 Boehringer Ingelheim Investigational Site, Charlotte, North Carolina
  - 1245.48.10005 Boehringer Ingelheim Investigational Site, Akron, Ohio
  - 1245.48.10004 Boehringer Ingelheim Investigational Site, Kettering, Ohio
  - 1245.48.10013 Boehringer Ingelheim Investigational Site, Erie, Pennsylvania
  - 1245.48.10020 Boehringer Ingelheim Investigational Site, Pittsburgh, Pennsylvania
  - 1245.48.10029 Boehringer Ingelheim Investigational Site, Knoxville, Tennessee
  - 1245.48.10015 Boehringer Ingelheim Investigational Site, Memphis, Tennessee
  - 1245.48.10034 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 1245.48.10007 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1245.48.10009 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1245.48.10042 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1245.48.10026 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 1245.48.10003 Boehringer Ingelheim Investigational Site, Orem, Utah
  - 1245.48.10023 Boehringer Ingelheim Investigational Site, Port Orchard, Washington
- Canada (7):
  - 1245.48.20002 Boehringer Ingelheim Investigational Site, Winnipeg, Manitoba
  - 1245.48.20001 Boehringer Ingelheim Investigational Site, Halifax, Nova Scotia
  - 1245.48.20004 Boehringer Ingelheim Investigational Site, Brampton, Ontario
  - 1245.48.20006 Boehringer Ingelheim Investigational Site, Etobicoke, Ontario
  - 1245.48.20007 Boehringer Ingelheim Investigational Site, Oakville, Ontario
  - 1245.48.20005 Boehringer Ingelheim Investigational Site, Thornhill, Ontario
  - 1245.48.20003 Boehringer Ingelheim Investigational Site, Toronto, Ontario
- Czechia (8):
  - 1245.48.42003 Boehringer Ingelheim Investigational Site, Benešov
  - 1245.48.42005 Boehringer Ingelheim Investigational Site, Brno
  - 1245.48.42002 Boehringer Ingelheim Investigational Site, Mladá Boleslav
  - 1245.48.42006 Boehringer Ingelheim Investigational Site, Neratovice
  - 1245.48.42008 Boehringer Ingelheim Investigational Site, Olomouc
  - 1245.48.42004 Boehringer Ingelheim Investigational Site, Opočno
  - 1245.48.42007 Boehringer Ingelheim Investigational Site, Příbram
  - 1245.48.42001 Boehringer Ingelheim Investigational Site, Slaný
- Denmark (10):
  - 1245.48.45006 Boehringer Ingelheim Investigational Site, Aalborg
  - 1245.48.45009 Boehringer Ingelheim Investigational Site, Aarhus C
  - 1245.48.45002 Boehringer Ingelheim Investigational Site, Elsinore
  - 1245.48.45008 Boehringer Ingelheim Investigational Site, Hellerup
  - 1245.48.45010 Boehringer Ingelheim Investigational Site, Hillerød
  - 1245.48.45003 Boehringer Ingelheim Investigational Site, København NV
  - 1245.48.45001 Boehringer Ingelheim Investigational Site, Rødovre Municipality
  - 1245.48.45004 Boehringer Ingelheim Investigational Site, Rødovre Municipality
  - 1245.48.45005 Boehringer Ingelheim Investigational Site, Vaerløse
  - 1245.48.45007 Boehringer Ingelheim Investigational Site, Vojens
- Estonia (4):
  - 1245.48.37203 Boehringer Ingelheim Investigational Site, Pärnu
  - 1245.48.37201 Boehringer Ingelheim Investigational Site, Tallinn
  - 1245.48.37202 Boehringer Ingelheim Investigational Site, Tallinn
  - 1245.48.37204 Boehringer Ingelheim Investigational Site, Tallinn
- Finland (7):
  - 1245.48.35802 Boehringer Ingelheim Investigational Site, Helsinki
  - 1245.48.35805 Boehringer Ingelheim Investigational Site, Joensuu
  - 1245.48.35806 Boehringer Ingelheim Investigational Site, Kouvola
  - 1245.48.35803 Boehringer Ingelheim Investigational Site, Oulu
  - 1245.48.35804 Boehringer Ingelheim Investigational Site, Pori
  - 1245.48.35801 Boehringer Ingelheim Investigational Site, Turku
  - 1245.48.35807 Boehringer Ingelheim Investigational Site, Turku
- France (7):
  - 1245.48.33004 Boehringer Ingelheim Investigational Site, Angers
  - 1245.48.33008 Boehringer Ingelheim Investigational Site, Bourges
  - 1245.48.33005 Boehringer Ingelheim Investigational Site, Mont-de-Marsan
  - 1245.48.33001 Boehringer Ingelheim Investigational Site, Nantes
  - 1245.48.33006 Boehringer Ingelheim Investigational Site, Orthez
  - 1245.48.33003 Boehringer Ingelheim Investigational Site, Tiercé
  - 1245.48.33007 Boehringer Ingelheim Investigational Site, Tours
- Germany (10):
  - 1245.48.49001 Boehringer Ingelheim Investigational Site, Berlin
  - 1245.48.49008 Boehringer Ingelheim Investigational Site, Berlin
  - 1245.48.49003 Boehringer Ingelheim Investigational Site, Dresden
  - 1245.48.49004 Boehringer Ingelheim Investigational Site, Hanover
  - 1245.48.49005 Boehringer Ingelheim Investigational Site, Lüneburg
  - 1245.48.49002 Boehringer Ingelheim Investigational Site, Mainz
  - 1245.48.49010 Boehringer Ingelheim Investigational Site, Nuremberg
  - 1245.48.49009 Boehringer Ingelheim Investigational Site, Pirna
  - 1245.48.49007 Boehringer Ingelheim Investigational Site, Schkeuditz
  - 1245.48.49006 Boehringer Ingelheim Investigational Site, Teuchern
- Lebanon (3):
  - 1245.48.96003 Boehringer Ingelheim Investigational Site, Baabda
  - 1245.48.96001 Boehringer Ingelheim Investigational Site, Beirut
  - 1245.48.96002 Boehringer Ingelheim Investigational Site, Lebanon
- Netherlands (14):
  - 1245.48.31011 Boehringer Ingelheim Investigational Site, Breda
  - 1245.48.31012 Boehringer Ingelheim Investigational Site, Eindhoven
  - 1245.48.31009 Boehringer Ingelheim Investigational Site, Etten-Leur
  - 1245.48.31014 Boehringer Ingelheim Investigational Site, Groningen
  - 1245.48.31013 Boehringer Ingelheim Investigational Site, Leiderdorp
  - 1245.48.31003 Boehringer Ingelheim Investigational Site, Oude Pekela
  - 1245.48.31016 Boehringer Ingelheim Investigational Site, Rotterdam
  - 1245.48.31006 Boehringer Ingelheim Investigational Site, Soerendonk
  - 1245.48.31008 Boehringer Ingelheim Investigational Site, Spijkenisse
  - 1245.48.31002 Boehringer Ingelheim Investigational Site, Swifterbant
  - 1245.48.31015 Boehringer Ingelheim Investigational Site, Velp
  - 1245.48.31010 Boehringer Ingelheim Investigational Site, Woerden
  - 1245.48.31019 Boehringer Ingelheim Investigational Site, Zijndrecht
  - 1245.48.31017 Boehringer Ingelheim Investigational Site, Zoetermeer
- Norway (9):
  - 1245.48.47009 Boehringer Ingelheim Investigational Site, Ålesund
  - 1245.48.47008 Boehringer Ingelheim Investigational Site, Elverum
  - 1245.48.47007 Boehringer Ingelheim Investigational Site, Hamar
  - 1245.48.47002 Boehringer Ingelheim Investigational Site, Kløfta
  - 1245.48.47001 Boehringer Ingelheim Investigational Site, Oslo
  - 1245.48.47003 Boehringer Ingelheim Investigational Site, Oslo
  - 1245.48.47004 Boehringer Ingelheim Investigational Site, Oslo
  - 1245.48.47005 Boehringer Ingelheim Investigational Site, Oslo
  - 1245.48.47006 Boehringer Ingelheim Investigational Site, Sørumsand
- Sweden (6):
  - 1245.48.46002 Boehringer Ingelheim Investigational Site, Härnösand
  - 1245.48.46004 Boehringer Ingelheim Investigational Site, Järfälla
  - 1245.48.46003 Boehringer Ingelheim Investigational Site, Lund
  - 1245.48.46007 Boehringer Ingelheim Investigational Site, Malmo
  - 1245.48.46006 Boehringer Ingelheim Investigational Site, Skene
  - 1245.48.46001 Boehringer Ingelheim Investigational Site, Stockholm

IPD SHARING:
Plan to Share IPD: Yes
Boehringer Ingelheim Policy on Transparency and Publication http://trials.boehringer-ingelheim.com/transparency_policy.html

REFERENCES:
- [Derived] Natale P, Tunnicliffe DJ, Toyama T, Palmer SC, Saglimbene VM, Ruospo M, Gargano L, Stallone G, Gesualdo L, Strippoli GF. Sodium-glucose co-transporter protein 2 (SGLT2) inhibitors for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 May 21;5(5):CD015588. doi: 10.1002/14651858.CD015588.pub2. PMID 38770818
- [Derived] Tuttle KR, Levin A, Nangaku M, Kadowaki T, Agarwal R, Hauske SJ, Elsasser A, Ritter I, Steubl D, Wanner C, Wheeler DC. Safety of Empagliflozin in Patients With Type 2 Diabetes and Chronic Kidney Disease: Pooled Analysis of Placebo-Controlled Clinical Trials. Diabetes Care. 2022 Jun 2;45(6):1445-1452. doi: 10.2337/dc21-2034. PMID 35472672
- [Derived] Mancia G, Cannon CP, Tikkanen I, Zeller C, Ley L, Woerle HJ, Broedl UC, Johansen OE. Impact of Empagliflozin on Blood Pressure in Patients With Type 2 Diabetes Mellitus and Hypertension by Background Antihypertensive Medication. Hypertension. 2016 Dec;68(6):1355-1364. doi: 10.1161/HYPERTENSIONAHA.116.07703. Epub 2016 Oct 10. PMID 27977392
- [Derived] Tikkanen I, Narko K, Zeller C, Green A, Salsali A, Broedl UC, Woerle HJ; EMPA-REG BP Investigators. Empagliflozin reduces blood pressure in patients with type 2 diabetes and hypertension. Diabetes Care. 2015 Mar;38(3):420-8. doi: 10.2337/dc14-1096. Epub 2014 Sep 30. PMID 25271206

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: A placebo tablet, matching the empagliflozin 10mg and 25mg tablets, taken once daily for 12 weeks.
- Empa 10mg: Single oral dose of empagliflozin (empa) 10mg taken once daily for 12 weeks.
- Empa 25mg: Single oral dose of empagliflozin (empa) 25mg taken once daily for 12 weeks.
Period: Overall Study
Arm/Group | Placebo | Empa 10mg | Empa 25mg
Started | 272 | 276 | 277
Completed | 256 | 265 | 266
Not Completed | 16 | 11 | 11
Not completed — Not treated | 1 | 0 | 0
Not completed — Adverse Event | 5 | 5 | 6
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — Non compliant with protocol | 0 | 1 | 2
Not completed — Lost to Follow-up | 1 | 1 | 1
Not completed — Patient refusal to continue,not due toAE | 5 | 4 | 0
Not completed — Other reason not defined above | 3 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomised and treated patients who had a baseline HbA1c value and a baseline mean 24-h SBP value. Treatment assignment as randomized
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Empa 10mg | Empa 25mg | Total
Number analyzed (Participants) | 271 | 276 | 276 | 823
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (8.8) | 60.6 (8.5) | 59.9 (9.7) | 60.2 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 105 | 120 | 328
  Male | 168 | 171 | 156 | 495

OUTCOME MEASURES:

1. Primary Outcome: HbA1c Change From Baseline
Description: Change from baseline in HbA1c after 12 weeks of treatment.
Time Frame: Baseline and 12 weeks
Population: Full analysis set (FAS), which included all randomised and treated patients who had a baseline HbA1c and a baseline mean 24-h systolic blood pressure value. Treatment assignment as randomised.
  Values after start of antidiabetic rescue therapy were set to missing and last observation carried forward (LOCF) was used for imputation of missing values.
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | Placebo | Empa 10mg | Empa 25mg
Number analyzed (Participants) | 271 | 276 | 276
percentage of HbA1c | 0.03 (0.60) | -0.59 (0.63) | -0.63 (0.62)
Statistical Analysis 1: Comparison: Placebo vs Empa 10mg; Hierarchical testing structure was: 1) Change from baseline to week 12 in HbA1c, empa 25mg vs placebo 2) Change from baseline to week 12 in mean 24h SBP, empa 25mg vs placebo 3) Change from baseline to week 12 in HbA1c, empa 10mg vs placebo 4) Change from baseline in mean 24h SBP, empa 10mg vs placebo 5) Change from baseline in mean 24h DBP, empa 25mg vs placebo 6) Change from baseline in mean 24h DBP empa 10mg vs placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — Hierarchical testing, no adjustment of p-values; Model includes baseline HbA1c as lin. covariate and treatment, baseline renal function, region and baseline N of antihyperten. med. as fixed effects; Mean Difference (Final Values) = -0.62, 95% CI 2-sided [-0.72 to -0.52], Standard Error of Mean 0.05 — Difference calculated as empa 10mg minus placebo
Statistical Analysis 2: Comparison: Placebo vs Empa 25mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — Hierarchical testing, no adjustment of p-values; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.65, 95% CI 2-sided [-0.75 to -0.55], Standard Error of Mean 0.05 — Difference calculated as empa 25mg minus placebo

2. Primary Outcome: Mean 24-hour Systolic Blood Pressure Change From Baseline
Description: Change from baseline of mean 24-hour systolic blood pressure (SBP).
Time Frame: Baseline and 12 weeks
Population: FAS, which included all randomised and treated patients who had a baseline HbA1c and a baseline mean 24-h systolic blood pressure value. Treatment assignment as randomised.
  Values after start of antidiabetic rescue therapy or change of antihypertensive therapy were set to missing and LOCF was used for imputation of missing values.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | Empa 10mg | Empa 25mg
Number analyzed (Participants) | 271 | 276 | 276
mmHg | 0.42 (8.25) | -2.99 (8.86) | -3.59 (9.30)
Statistical Analysis 1: Comparison: Placebo vs Empa 10mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — Hierarchical testing, no adjustment of p-values; Model incl. baseline (bl) HbA1c, bl mean 24h SBP as lin. covariates; treatment, bl renal function, region, bl N of antihyperten. med. as fixed effects; Mean Difference (Final Values) = -3.44, 95% CI 2-sided [-4.78 to -2.09], Standard Error of Mean 0.69 — Difference calculated as empa 10mg minus placebo
Statistical Analysis 2: Comparison: Placebo vs Empa 25mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — Hierarchical testing, no adjustment of p-values; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -4.16, 95% CI 2-sided [-5.50 to -2.83], Standard Error of Mean 0.68 — Difference calculated as empa 25mg minus placebo

3. Secondary Outcome: Mean 24-hour Diastolic Blood Pressure Change From Baseline
Description: Change from baseline in mean 24-hour diastolic blood pressure (DBP) after 12 weeks.
Time Frame: Baseline and 12 weeks
Population: FAS which included all randomised and treated patients who had a baseline HbA1c and a baseline mean 24-h systolic blood pressure value. Treatment assignment as randomised.
  Values after start of antidiabetic rescue therapy or change of antihypertensive therapy were set to missing and LOCF was used for imputation of missing values.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | Empa 10mg | Empa 25mg
Number analyzed (Participants) | 271 | 276 | 276
mmHg | 0.30 (5.06) | -1.10 (4.96) | -1.32 (4.96)
Statistical Analysis 1: Comparison: Placebo vs Empa 10mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0008, ANCOVA — Hierarchical testing, no adjustment of p-values; Model incl. baseline (bl) HbA1c, bl mean 24h DBP as lin. covariates; treatment, bl renal function, region, bl N of antihyperten. med. as fixed effects; Mean Difference (Final Values) = -1.36, 95% CI 2-sided [-2.15 to -0.56], Standard Error of Mean 0.40 — Difference calculated as empa 10mg minus placebo
Statistical Analysis 2: Comparison: Placebo vs Empa 25mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — Hierarchical testing, no adjustment of p-values; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = -1.72, 95% CI 2-sided [-2.51 to -0.93], Standard Error of Mean 0.40 — Difference calculated as empa 25mg minus placebo

4. Secondary Outcome: Proportion of Patients With HbA1c <7%
Description: Proportion of patients with HbA1c <7% after 12 weeks.
Time Frame: Baseline and 12 weeks
Population: Patients in the full analysis set (FAS) and with baseline HbA1c >= 7%. Treatment assignment as randomised.
  Non-completers (missing data due to early discontinuation or values after start of rescue medication) considered 'failure' was used as the imputation rule.
Measure: Number; unit: participants
Arm/Group | Placebo | Empa 10mg | Empa 25mg
Number analyzed (Participants) | 252 | 256 | 264
participants | 18 | 79 | 79
Statistical Analysis 1: Comparison: Placebo vs Empa 10mg; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Logistic regression model includes treatment, baseline renal function, region, baseline number of antihypertensive medications and baseline HbA1c; Odds Ratio (OR) = 6.26, 95% CI 2-sided [3.51 to 11.18]
Statistical Analysis 2: Comparison: Placebo vs Empa 25mg; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; [statistical method as in outcome 4, analysis 1]; Odds Ratio (OR) = 6.59, 95% CI 2-sided [3.70 to 11.75]

5. Secondary Outcome: Fasting Plasma Glucose (FPG) Change From Baseline
Description: Change from baseline in FPG after 12 weeks of treatment.
Time Frame: Baseline and 12 weeks
Population: Full analysis set (FAS) which included all randomised and treated patients who had a baseline HbA1c value and a baseline mean 24-h systolic blood pressure (SBP) value. Treatment assignment as randomised.
  Values after start of antidiabetic rescue therapy were set to missing and LOCF was used for imputation of missing values.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Empa 10mg | Empa 25mg
Number analyzed (Participants) | 271 | 276 | 276
mg/dL | 7.19 (38.29) | -15.23 (33.32) | -24.45 (35.38)
Statistical Analysis 1: Comparison: Placebo vs Empa 10mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Model includes treatment, baseline renal function, geographical region, baseline N of antihyperten. med., baseline HbA1c and baseline FPG; Mean Difference (Final Values) = -23.76, 95% CI 2-sided [-28.91 to -18.60], Standard Error of Mean 2.63 — Difference calculated as empa 10mg minus placebo
Statistical Analysis 2: Comparison: Placebo vs Empa 25mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -30.20, 95% CI 2-sided [-35.32 to -25.08], Standard Error of Mean 2.61 — Difference calculated as empa 25mg minus placebo

6. Secondary Outcome: Body Weight Change From Baseline
Description: Change from baseline in body weight after 12 weeks of treatment.
Time Frame: Baseline and 12 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Placebo | Empa 10mg | Empa 25mg
Number analyzed (Participants) | 271 | 276 | 276
kg | -0.19 (1.55) | -1.67 (2.38) | -2.16 (2.38)
Statistical Analysis 1: Comparison: Placebo vs Empa 10mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Model includes treatment, baseline renal function, geographical region, baseline number of antihypertensive med., baseline HbA1c and baseline weight; Mean Difference (Final Values) = -1.49, 95% CI 2-sided [-1.85 to -1.13], Standard Error of Mean 0.18 — Difference calculated as empa 10mg minus placebo
Statistical Analysis 2: Comparison: Placebo vs Empa 25mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 6, analysis 1]; Mean Difference (Final Values) = -1.98, 95% CI 2-sided [-2.33 to -1.62], Standard Error of Mean 0.18 — Difference calculated as empa 10mg minus placebo

7. Secondary Outcome: Daytime Mean Systolic Blood Pressure (SBP) Change From Baseline
Description: Change from baseline in daytime mean SBP after 12 weeks of treatment.
Time Frame: Baseline and 12 weeks
Population: FAS which included all randomised and treated patients who had a baseline HbA1c value and a baseline mean 24-h systolic blood pressure (SBP) value. Treatment assignment as randomised.
  Values after start of antidiabetic rescue therapy or change of antihypertensive therapy were set to missing and LOCF was used for imputation of missing values.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | Empa 10mg | Empa 25mg
Number analyzed (Participants) | 271 | 276 | 276
mmHg | 0.38 (8.74) | -3.40 (9.55) | -4.12 (9.55)
Statistical Analysis 1: Comparison: Placebo vs Empa 10mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Model includes treatment, baseline renal function, geographical region, N of antihypertensive medications, baseline HbA1c and baseline daytime SBP; Mean Difference (Final Values) = -3.94, 95% CI 2-sided [-5.37 to -2.52], Standard Error of Mean 0.73 — Difference calculated as empa 10mg minus placebo
Statistical Analysis 2: Comparison: Placebo vs Empa 25mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Model includes treatment, baseline renal function, geographical region, baseline N of antihyperten. med., baseline HbA1c and baseline daytime SBP; Mean Difference (Final Values) = -4.78, 95% CI 2-sided [-6.20 to -3.36], Standard Error of Mean 0.72 — Difference calculated as empa 25mg minus placebo

8. Secondary Outcome: Daytime Mean Diastolic Blood Pressure (DBP) Change From Baseline
Description: Change from baseline in daytime mean DBP after 12 weeks of treatment.
Time Frame: Baseline and 12 weeks
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | Empa 10mg | Empa 25mg
Number analyzed (Participants) | 271 | 276 | 276
mmHg | 0.26 (5.36) | -1.28 (5.41) | -1.58 (5.35)
Statistical Analysis 1: Comparison: Placebo vs Empa 10mg; Test type: Superiority or Other; p = 0.0004, ANCOVA; Model includes treatment, baseline renal function, geographical region, baseline N of antihyperten. med., baseline HbA1c and baseline daytime DBP; Mean Difference (Final Values) = -1.56, 95% CI 2-sided [-2.42 to -0.69], Standard Error of Mean 0.44 — Difference calculated as empa 10mg minus placebo
Statistical Analysis 2: Comparison: Placebo vs Empa 25mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 8, analysis 1]; Mean Difference (Final Values) = -1.98, 95% CI 2-sided [-2.84 to -1.12], Standard Error of Mean 0.44 — Difference calculated as empa 25mg minus placebo

9. Secondary Outcome: Nighttime Mean Systolic Blood Pressure (SBP) Change From Baseline
Description: Change from baseline in nighttime mean SBP after 12 weeks of treatment.
Time Frame: Baseline and 12 weeks
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | Empa 10mg | Empa 25mg
Number analyzed (Participants) | 271 | 276 | 276
mmHg | 0.51 (10.22) | -2.22 (10.21) | -2.47 (11.09)
Statistical Analysis 1: Comparison: Placebo vs Empa 10mg; Test type: Superiority or Other; p = 0.0021, ANCOVA; Model includes treatment, baseline renal function, geographical region, baseline N of antihyperten. med., baseline HbA1c and baseline night-time SBP; Mean Difference (Final Values) = -2.50, 95% CI 2-sided [-4.09 to -0.91], Standard Error of Mean 0.81 — Difference calculated as empa 10mg minus placebo
Statistical Analysis 2: Comparison: Placebo vs Empa 25mg; Test type: Superiority or Other; p = 0.0003, ANCOVA; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -2.90, 95% CI 2-sided [-4.48 to -1.32], Standard Error of Mean 0.81 — Difference calculated as empa 25mg minus placebo

10. Secondary Outcome: Nighttime Mean Diastolic Blood Pressure (DBP) Change From Baseline
Description: Change from baseline in nighttime mean DBP after 12 weeks of treatment.
Time Frame: Baseline and 12 weeks
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | Empa 10mg | Empa 25mg
Number analyzed (Participants) | 271 | 276 | 276
mmHg | 0.36 (6.80) | -0.80 (6.21) | -0.75 (6.32)
Statistical Analysis 1: Comparison: Placebo vs Empa 10mg; Test type: Superiority or Other; p = 0.0566, ANCOVA; Model includes treatment, baseline renal function, geographical region, baseline N of antihyperten. med., baseline HbA1c and baseline night-time DBP; Mean Difference (Final Values) = -0.95, 95% CI 2-sided [-1.93 to 0.03], Standard Error of Mean 0.50 — Difference calculated as empa 10mg minus placebo
Statistical Analysis 2: Comparison: Placebo vs Empa 25mg; Test type: Superiority or Other; p = 0.0208, ANCOVA; [statistical method as in outcome 10, analysis 1]; Mean Difference (Final Values) = -1.15, 95% CI 2-sided [-2.12 to -0.18], Standard Error of Mean 0.50 — Difference calculated as empa 25mg minus placebo

11. Secondary Outcome: Trough Mean Seated Systolic Blood Pressure (SBP) Change From Baseline
Description: Change from baseline in Trough Mean Seated SBP after 12 weeks of treatment.
Time Frame: Baseline and 12 weeks
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | Empa 10mg | Empa 25mg
Number analyzed (Participants) | 271 | 276 | 276
mmHg | -0.57 (11.92) | -4.73 (12.54) | -5.45 (12.43)
Statistical Analysis 1: Comparison: Placebo vs Empa 10mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Model includes treatment, baseline renal function, geographical region, baseline N of antihyperten. med., baseline HbA1c and baseline seated SBP; Mean Difference (Final Values) = -3.92, 95% CI 2-sided [-5.86 to -1.98], Standard Error of Mean 0.99 — Difference calculated as empa 10mg minus placebo
Statistical Analysis 2: Comparison: Placebo vs Empa 25mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 11, analysis 1]; Mean Difference (Final Values) = -4.80, 95% CI 2-sided [-6.73 to -2.87], Standard Error of Mean 0.98 — Difference calculated as empa 25mg minus placebo

12. Secondary Outcome: Trough Mean Seated Diastolic Blood Pressure (DBP) Change From Baseline
Description: Change from baseline in trough mean seated DBP after 12 weeks of treatment.
Time Frame: Baseline and 12 weeks
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | Empa 10mg | Empa 25mg
Number analyzed (Participants) | 271 | 276 | 276
mmHg | -1.02 (6.58) | -3.18 (7.10) | -3.01 (7.05)
Statistical Analysis 1: Comparison: Placebo vs Empa 10mg; Test type: Superiority or Other; p = 0.0005, ANCOVA; Model includes treatment, baseline renal function, geographical region, baseline N of antihyperten. med., baseline HbA1c and baseline seated DBP; Mean Difference (Final Values) = -1.93, 95% CI 2-sided [-3.01 to -0.84], Standard Error of Mean 0.55 — Difference calculated as empa 10mg minus placebo
Statistical Analysis 2: Comparison: Placebo vs Empa 25mg; Test type: Superiority or Other; p = 0.0006, ANCOVA; [statistical method as in outcome 12, analysis 1]; Mean Difference (Final Values) = -1.89, 95% CI 2-sided [-2.97 to -0.82], Standard Error of Mean 0.55 — Difference calculated as empa 25mg minus placebo

13. Secondary Outcome: Proportion of Patients Reaching Blood Pressure <130/80 mmHg
Description: Proportion of patients reaching blood pressure <130/80 mmHg after 12 weeks of treatment
Time Frame: Baseline and 12 weeks
Population: Patients in the FAS without blood pressure control at baseline. Blood pressure control is defined as DBP<80 mmHg and SBP <130 mmHg. Treatment assignment as randomised.
  Non-completers (missing data due to early disc, values after start of rescue medication or changes in antihyp. therapy) considered 'failure' was used as the imputation rule.
Measure: Number; unit: participants
Arm/Group | Placebo | Empa 10mg | Empa 25mg
Number analyzed (Participants) | 241 | 251 | 247
participants | 19 | 45 | 40
Statistical Analysis 1: Comparison: Placebo vs Empa 10mg; Test type: Superiority or Other; p = 0.0021, Regression, Logistic; [statistical method as in outcome 4, analysis 1]; Odds Ratio (OR) = 2.49, 95% CI 2-sided [1.39 to 4.45]
Statistical Analysis 2: Comparison: Placebo vs Empa 25mg; Test type: Superiority or Other; p = 0.0088, Regression, Logistic; [statistical method as in outcome 4, analysis 1]; Odds Ratio (OR) = 2.20, 95% CI 2-sided [1.22 to 3.96]

14. Secondary Outcome: Composite Endpoint of Change From Baseline of HbA1c, Systolic Blood Pressure and Body Weight
Description: A composite endpoint of the following conditions at week 12 compared to baseline (all 3 fulfilled): reduction of HbA1c from baseline of at least 0.5%, reduction of systolic blood pressure > 3 mmHg from baseline and reduction of weight from baseline > 2%
Time Frame: Baseline and 12 weeks
Population: Patients in the full analysis set (FAS). Treatment assignment as randomised.
  Non-completers (missing data due to early discontinuation, values after start of rescue medication or changes in antihypertensive therapy) considered 'failure' was used as the imputation rule.
Measure: Number; unit: participants
Arm/Group | Placebo | Empa 10mg | Empa 25mg
Number analyzed (Participants) | 271 | 276 | 276
participants
  Number fulfilled | 6 | 41 | 58
  Number not fulfilled | 265 | 235 | 218

15. Secondary Outcome: Orthostatic Blood Pressure
Description: Orthostatic blood pressure (BP) at baseline and after 12 weeks of treatment.
Time Frame: Baseline and 12 weeks
Population: Treated set for patients with available measurements at baseline and week 12. Treatment assignment as first medication taken.
Measure: Number; unit: participants
Arm/Group | Placebo | Empa 10mg | Empa 25mg
Number analyzed (Participants) | 254 | 259 | 259
participants
  Baseline: Positive | 42 | 40 | 51
  Baseline: Negative | 212 | 219 | 208
  Week 12: Positive | 51 | 67 | 76
  Week 12: Negative | 203 | 192 | 183

16. Other Pre Specified Outcome: Confirmed Hypoglycaemic Adverse Events
Description: Number of participants with confirmed hypoglycaemic adverse events
Time Frame: From drug administration until last drug administration plus seven days, up to 171 days
Population: Treated set which included all patients treated with at least one dose of randomised trial medication. Treatment assignment as first medication taken.
Measure: Number; unit: participants
Arm/Group | Placebo | Empa 10mg | Empa 25mg
Number analyzed (Participants) | 272 | 276 | 276
participants | 13 | 18 | 17

ADVERSE EVENTS:
Time Frame: From drug administration until last drug administration plus seven days, up to 171 days
Arm/Group | Placebo | Empa 10mg | Empa 25mg
Serious Adverse Events (participants affected / at risk) | 7/272 | 3/276 | 4/276
Other Adverse Events (participants affected / at risk) | 43/272 | 42/276 | 55/276
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=272) | Empa 10mg (N=276) | Empa 25mg (N=276)
Osteomyelitis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Carotid artery thrombosis (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0
Acute vestibular syndrome (Ear and labyrinth disorders) | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Urethral stenosis (Renal and urinary disorders) | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1
Sudden death (General disorders) | 0 | 1 | 0
Electrocardiogram T wave inversion (Investigations) | 0 | 0 | 1
Traumatic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=272) | Empa 10mg (N=276) | Empa 25mg (N=276)
Nasopharyngitis (Infections and infestations) | 26 | 15 | 20
Hypoglycaemia (Metabolism and nutrition disorders) | 14 | 19 | 19
Pollakiuria (Renal and urinary disorders) | 7 | 11 | 17
Thirst (General disorders) | 1 | 2 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.